CLINICAL TRIAL: NCT02446405
Title: Randomised Phase 3 Trial of Enzalutamide in First Line Androgen Deprivation Therapy for Metastatic Prostate Cancer: ENZAMET
Brief Title: Enzalutamide in First Line Androgen Deprivation Therapy for Metastatic Prostate Cancer
Acronym: ENZAMET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Cancer Trials Ireland (Network); Canadian Cancer Trials Group (Network); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1304; ACTRN12614000110684 (Other: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2015-05-04; First posted 2015-05-18 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Neoplasms
Keywords: metastatic prostate cancer; prostate cancer; prostate cancer treatment; enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Castration

STUDY DESIGN:
Intervention Model Description: Stratification factors:
  1. High volume disease (yes versus no), characterised as:
     * 4 or more bone metastases, one of which is outside the vertebral column and pelvis AND/OR
     * Visceral metastases (e.g. lung, pleura, liver, adrenal and others) Lymph node involvement or bladder invasion do NOT qualify as visceral disease.
  2. Study site
  3. Concomitant "anti-resorptive" therapy to delay skeletal related events when commencing ADT
  4. Co-morbidities according to the Adult Co-morbidity Evaluation (ACE-27: 0-1 vs 2-3)
  5. Early use of docetaxel defined as use of docetaxel in conjunction with initiation of ADT.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzalutamide (Experimental): Enzalutamide is 160 mg daily, by mouth, until clinical disease progression or prohibitive toxicity.
  All participants are to receive standard background therapy with a LHRHA or surgical castration, as per standard of care. The choice of the LHRHA or surgical castration is at the discretion of the treating clinician.
  Interventions: Drug: Enzalutamide; Drug: LHRHA or Surgical Castration
- Conventional NSAA (Active Comparator): Conventional NSAA, by mouth until clinical disease progression or prohibitive toxicity.
  All participants are to receive standard background therapy with a LHRHA or surgical castration, as per standard of care. The choice of the LHRHA or surgical castration is at the discretion of the treating clinician.
  Interventions: Drug: NSAA; Drug: LHRHA or Surgical Castration

INTERVENTIONS:
Drug: Enzalutamide
  Arms: Enzalutamide
Drug: NSAA
  Arms: Conventional NSAA
Drug: LHRHA or Surgical Castration

SUMMARY:
The purpose of this study is to determine the effectiveness of enzalutamide, versus a conventional non-steroidal anti androgen (NSAA), when combined with a luteinizing hormone releasing hormone analog (LHRHA) or surgical castration, as first line androgen deprivation therapy (ADT) for newly diagnosed metastatic prostate cancer.

ELIGIBILITY:
Men starting first line androgen deprivation therapy for metastatic prostate cancer.

Inclusion criteria:

1. Male aged 18 or older with metastatic adenocarcinoma of the prostate
2. Target or non-target lesions according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1
3. Adequate bone marrow function: Haemoglobin (Hb) ≥100g/L and White Cell Count (WCC) ≥ 4.0 x 109/L and platelets ≥100 x 109/L.
4. Adequate liver function: Alanine transaminase (ALT) < 2 x Upper Limit of Normal (ULN) and bilirubin < 1.5 x ULN, (or if bilirubin is between 1.5-2 x ULN, they must have a normal conjugated bilirubin). If liver metastases are present ALT must be < 5 x ULN
5. Adequate renal function: calculated creatinine clearance > 30 ml/min (Cockcroft-Gault)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. Patients with performance status 2 are only eligible if the decline in performance status is due to metastatic prostate cancer.
7. Study treatment both planned and able to start within 7 days after randomisation.
8. Willing and able to comply with all study requirements, including treatment and required assessments
9. Has completed baseline Health-Related Quality of Life (HRQL) questionnaires UNLESS is unable to complete because of limited literacy or vision
10. Signed, written, informed consent

Exclusion Criteria:

1. Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components
2. History of

   * seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma).
   * loss of consciousness or transient ischemic attack within 12 months of randomization
   * significant cardiovascular disease within the last 3 months including: myocardial infarction, unstable angina, congestive heart failure, ongoing arrhythmias of Grade >2 [National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.03], thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism). Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
3. Life expectancy of less than 12 months.
4. History of another malignancy within 5 years prior to randomisation, except for either non- melanomatous carcinoma of the skin or, adequately treated, non-muscle-invasive urothelial carcinoma of the bladder (Tis, Ta and low grade T1 tumours).
5. Concurrent illness, including severe infection that might jeopardize the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety

   a. Human Immunodeficiency Virus (HIV)-infection is not an exclusion criterion if it is controlled with anti-retroviral drugs that are unaffected by concomitant enzalutamide.
6. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse;
7. Patients who are sexually active and not willing/able to use medically acceptable forms of barrier contraception.
8. Prior ADT for prostate cancer (including bilateral orchidectomy), except in the following settings:

   * Started less than 12 weeks prior to randomisation AND Prostate Specific Antigen (PSA) is stable or falling. The 12 weeks starts from whichever of the following occurs earliest: first dose of oral anti- androgen, LHRHA, or surgical castration.
   * In the adjuvant setting, where the completion of adjuvant hormonal therapy was more than 12 months prior to randomisation AND the total duration of hormonal treatment did not exceed 24 months. For depot preparations, hormonal therapy is deemed to have started with the first dose and to have been completed when the next dose would otherwise have been due, e.g. 12 weeks after the last dose of depot goserelin 10.8mg.
9. Prior cytotoxic chemotherapy for prostate cancer, but up to 2 cycles of docetaxel chemotherapy for metastatic disease is permitted.
10. Participation in other clinical trials of investigational agents for the treatment of prostate cancer or other diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1125 (Actual)
Dates: Start 2014-03; Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Time | 3 years
  the interval from the date of randomisation to date of death.

SECONDARY OUTCOMES:
Prostate specific antigen progression free survival time | 3 years
  the interval from the date of randomisation to the date of first evidence of PSA progression, clinical progression, or death from any cause, whichever occurs first, or the date of last known follow-up without PSA progression
  PSA progression is defined as: a rise in PSA by more than 25% AND more than 2ng/mL
Clinical progression free survival time | 3 years
  the interval from the date of randomisation to the date of first clinical evidence of disease progression or death from any cause, whichever occurs first, or the date of last known follow-up without clinical progression
Adverse events | 3 years
  The NCI Common Terminology Criteria for Adverse Events version 4 (CTCAE v4.03) will be used to classify and grade the intensity of adverse events during study treatment
Health-related quality of life (EORTC Core Quality of Life Questionnaire (QLQ C-30), Quality of Life Questionnaire for Prostate Cancer (PR-25), Euroqol 5 item preference-based measure of health (EQ-5 D-5L)) | 3 years
  HRQL will be reported by participants using the EORTC core quality of life questionnaire (QLQ C-30) and prostate cancer specific module (PR-25). The EQ-5D-5L will be used to derive utility scores suitable for quality adjusted survival analyses
Healthcare resource cost-effectiveness (incremental cost effectiveness ratio) | 3 years
  Information on the following areas of health-care resource usage will be collected: hospitalisations, visits to health professionals, and medications Australian unit costs will be applied to the resource usage data to estimate the incremental cost of the addition of enzalutamide to standard treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, Study Chair — Dana Farber Cancer Institute and ANZUP; Ian Davis, Study Chair — ANZUP and Eastern Health Box Hill Hospital
Locations (82):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States
- Australia (38):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Concord Cancer Centre - Concord Repatriation General Hospital, Concord, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Cancer Care Centre, Kingswood, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Central West Cancer Services, Orange, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Genesis Care North Shore, St Leonards, New South Wales
  - Tamworth Rural Referral Hospital, Tamworth, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Adelaide Cancer Centre - Ashford Cancer Care Centre, Kurralta Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Hospital, Bendigo, Victoria
  - Monash Cancer Centre Moorabbin, Bentleigh East, Victoria
  - Peter MacCallum Cancer Centre - East Melbourne, East Melbourne, Victoria
  - St. Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula South Eastern Haematology & Oncology Group- Peninsula Oncology Centre, Frankston, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Australian Urology Associates, Malvern, Victoria
  - Eastern Health Box Hill Hospital, Melbourne, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Fiona Stanley Hospital (formerly Royal Perth Hospital), Perth, Western Australia
- Canada (21):
  - Prostate Cancer Institute - Southern Alberta Institute of Urology, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Center, Surrey, British Columbia
  - BCCA Vancouver Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Horizon Health Network - Dr Everett Chalmers Hospital, Fredericton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre, Capital District Health Authority, Halifax, Nova Scotia
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - University Health Network - Princess Margaret Hospital, Toronto, Ontario
  - Hôpital Notre-Dame, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Ireland (9):
  - Beaumont Hospital, Beaumont, Dublin
  - Beacon Private Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Mater Misercordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James Hospital, Dublin
  - Galway University Hospital, Galway
  - Adelaide and Meath Hospital - National Children's Hospital, Tallaght
  - University Hospital Waterford, Waterford
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- United Kingdom (10):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Sussex Hospital, Brighton, East Sussex
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Velindre Cancer Centre, Cardiff, Wales
  - University College Hospital London, London
  - Guys and St Thomas Hospital, London
  - Royal Marsden Hospital, London
  - University Hospital Southampton, Southampton
  - Great Western Hospital, Swindon

REFERENCES:
- [Derived] Armstrong AJ, Azad AA, Conduit C, Haas GP, Bland C, Davis ID. Enzalutamide in metastatic hormone-sensitive prostate cancer: A plain language summary of the ARCHES and ENZAMET follow-up studies. Future Oncol. 2025 Jan;21(1):15-24. doi: 10.1080/14796694.2024.2408101. Epub 2024 Oct 15. PMID 39404227
- [Derived] Sweeney CJ, Martin AJ, Stockler MR, Begbie S, Cheung L, Chi KN, Chowdhury S, Frydenberg M, Horvath LG, Joshua AM, Lawrence NJ, Marx G, McCaffrey J, McDermott R, McJannett M, North SA, Parnis F, Parulekar W, Pook DW, Reaume MN, Sandhu SK, Tan A, Tan TH, Thomson A, Vera-Badillo F, Williams SG, Winter D, Yip S, Zhang AY, Zielinski RR, Davis ID; ENZAMET trial investigators and Australian and New Zealand Urogenital and Prostate Cancer Trials Group. Testosterone suppression plus enzalutamide versus testosterone suppression plus standard antiandrogen therapy for metastatic hormone-sensitive prostate cancer (ENZAMET): an international, open-label, randomised, phase 3 trial. Lancet Oncol. 2023 Apr;24(4):323-334. doi: 10.1016/S1470-2045(23)00063-3. PMID 36990608
- [Derived] Stockler MR, Martin AJ, Davis ID, Dhillon HM, Begbie SD, Chi KN, Chowdhury S, Coskinas X, Frydenberg M, Hague WE, Horvath LG, Joshua AM, Lawrence NJ, Marx GM, McCaffrey J, McDermott R, McJannett M, North SA, Parnis F, Parulekar WR, Pook DW, Reaume MN, Sandhu S, Tan A, Tan TH, Thomson A, Vera-Badillo F, Williams SG, Winter DG, Yip S, Zhang AY, Zielinski RR, Sweeney CJ; ENZAMET Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group (ANZUP). Health-Related Quality of Life in Metastatic, Hormone-Sensitive Prostate Cancer: ENZAMET (ANZUP 1304), an International, Randomized Phase III Trial Led by ANZUP. J Clin Oncol. 2022 Mar 10;40(8):837-846. doi: 10.1200/JCO.21.00941. Epub 2021 Dec 20. PMID 34928708
- [Derived] Davis ID, Martin AJ, Stockler MR, Begbie S, Chi KN, Chowdhury S, Coskinas X, Frydenberg M, Hague WE, Horvath LG, Joshua AM, Lawrence NJ, Marx G, McCaffrey J, McDermott R, McJannett M, North SA, Parnis F, Parulekar W, Pook DW, Reaume MN, Sandhu SK, Tan A, Tan TH, Thomson A, Tu E, Vera-Badillo F, Williams SG, Yip S, Zhang AY, Zielinski RR, Sweeney CJ; ENZAMET Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. Enzalutamide with Standard First-Line Therapy in Metastatic Prostate Cancer. N Engl J Med. 2019 Jul 11;381(2):121-131. doi: 10.1056/NEJMoa1903835. Epub 2019 Jun 2. PMID 31157964
- [Derived] Davis ID. Answering Questions and Questioning Answers: More Evidence To Guide Decision-making About Chemohormonal Therapy in Metastatic Prostate Cancer. Eur Urol. 2018 Jun;73(6):856-858. doi: 10.1016/j.eururo.2018.02.020. Epub 2018 Mar 7. No abstract available. PMID 29525541
- See also: Australian and New Zealand Urogenital and Prostate (ANZUP) Cancer Trials Group. — https://www.anzup.org.au/
- See also: University of Sydney, National Health and Medical Research Council (NHMRC) Clinical Trials Centre. — http://ctc.usyd.edu.au/
- See also: Australian New Zealand Clinical Trials Registry (ANZCTR) — http://www.anzctr.org.au/